CLINICAL TRIAL: NCT00221637
Title: Efficacy of a Therapeutic Strategy in Peripheral Neuropathic Pain: Intravenous Sodium Valproate Followed by Oral Route Treatment Versus Placebo (Clinical and Neurophysiologic Evaluation)
Brief Title: Efficacy of Valproate in Peripheral Neuropathic Pain
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: slow recruitment and treatments beyond expiry date
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9236-01; 2000-003
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Neuralgia; Neuropathic Peripheral Pain
Keywords: Neuralgia; Valproate; Anticonvulsant Drugs; Pain Measurement; Randomized Controlled Trials
MeSH Terms: conditions — Neuralgia | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sodium Valproate

SUMMARY:
The purpose of this study is to determine whether valproate is effective and well tolerated in the treatment of neuropathic peripheral pain. The drug is administered by intravenous route followed by oral route during 4 weeks.

DETAILED DESCRIPTION:
Background. Neuropathic peripheral pain is often refractory to usual analgesics. Some anticonvulsant drugs may be effective, but often partially only, and not always well tolerated. Valproate is a well-known anticonvulsant drug, with moderate possible adverse events and for which an intravenous form is available.

Aim. The principal aim is to assess the efficacy and safety of sodium Valproate in peripheral neuropathic pain. Secondary aims are to asses the effect of IV and oral treatment on neurophysiologic measures.

Design. Randomized, double-blind vs. placebo, parallel groups, monocentric clinical trial.

Treatments. Experimental arm: Intravenous eight-hour sodium Valproate infusion, followed by a four-week oral route sodium Valproate treatment. Control arm: Intravenous eight-hour placebo infusion, followed by a four-week oral route placebo treatment. Rescue medications are allowed in both groups.

Eligibility criteria. Peripheral neuropathic pain with pain intensity of at least 40 mm on a visual analog scale.

Outcomes. Primary outcome is the intensity of pain on a visual analog scale after 4 weeks of treatment. Secondary outcomes: intensity of pain after IV treatment; neurophysiologic measures (thermal thresholds, RIII reflex); association of response to IV treatment with oral treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* peripheral neuropathic pain
* signed written informed consent

Exclusion Criteria:

* central neuropathic pain
* current or past hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-03; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Intensity of pain on a visual analog scale | after 4 weeks of treatment

SECONDARY OUTCOMES:
intensity of mechanic allodynia
intensity of dynamic allodynia
use of analgesics (rescue medication)
thermal sensitive and nociceptive thresholds, RIII reflex

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Dousset, Dr, Principal Investigator — University Hospital, Bordeaux; Paul Perez, Dr, Study Chair — University Hospital, Bordeaux
Locations (1):
- Unité de traitement de la douleur chronique, Hôpital Pellegrin, CHU de Bordeaux, Bordeaux, France